CLINICAL TRIAL: NCT05663567
Title: TheEffect of a Solution-FocusedApproach on Breastfeeding Self-efficacy: A RandomizedControlledStudy
Brief Title: TheEffect of a Solution-FocusedApproach on Breastfeeding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, ESRA NUR KABAKCI, RESEARCH ASSİSTMENT, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SFAB
Record Dates: First submitted 2022-10-26; First posted 2022-12-23 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Postpartum; Breastfeeding; Self Efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group 1 (Experimental): Implementing a solution-focused approach to support breastfeeding ONE TO ONE STUDY
  Interventions: Behavioral: solution oriented approach
- experimental group 2 (Experimental): Implementing a solution-focused approach to support breastfeeding GROUP STUDY
  Interventions: Behavioral: solution oriented approach
- No Intervention (No Intervention): ROUTINE MAINTENANCE WILL BE DONE SOLUTION-FOCUSED APPROACH WILL NOT BE APPLIED.

INTERVENTIONS:
Behavioral: solution oriented approach — Implementing a solution-focused approach to support breastfeeding
  Arms: experimental group 1; experimental group 2

SUMMARY:
The Effect of a Solution-FocusedApproach on Breastfeeding Self-efficacy:

A RandomizedControlledStudy It is a single-blind, randomized controlled study with a pre-test post-test design.

In this study, it is aimed to increase the psychosocial health levels of mothers in the postpartum period and to eliminate their concerns about breastfeeding and infant feeding, with a solution-oriented approach planned to be applied to mothers with low breastfeeding self-efficacy. In addition, it is thought that the results of the research will make an important contribution to the national literature.

Question 1: Is a solution-oriented approach effective in increasing mothers' breastfeeding self-efficacy?

DETAILED DESCRIPTION:
Solution-Focused Approach (COS) is a therapeutic counseling method developed by Steve de Shazer and Insoo Kim Berg et al. in the mid-1970s. This postmodern approach method focuses on the solution itself rather than going to the root of the problems, revealing the individual's past achievements and positive experiences. aims to remove.

One of the most important advantages of the Solution-Oriented Approach is that it is effective in a short time. Studies have shown that CFS can achieve the desired results between 6 and 10 sessions. It is important that the sessions and techniques of the Solution-Oriented Approach are used in harmony and that the sessions are structured. Particular attention is paid to the first session as it initiates the change and contributes to the process. In Solution-Oriented Approach, sessions are conducted as "first session" and "second and other sessions".

In this study, it is aimed to increase the psychosocial health levels of mothers in the postpartum period and to eliminate their concerns about breastfeeding and infant feeding, with a solution-oriented approach planned to be applied to mothers with low breastfeeding self-efficacy. In addition, it is thought that the results of the research will make an important contribution to the national literature

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old, literate,
* Can speak Turkish,
* Primiparous and at term and healthy delivery (38-42 weeks, 2500-4000g born, 5th minute APGAR score of 7 and above, no known congenital disease),
* Women who do not have a chronic disease that prevents breastfeeding in their baby or in themselves
* Does not have a systemic disease,
* Those who have never received a planned breastfeeding training before,
* Having a healthy pregnancy,
* Planning to breastfeed,
* Women who have internet access, devices with internet usage (smartphone, computer, tablet, etc.), who have Zoom and Google Meet video conferencing applications on these devices.
* Women who can be reached within one week at the latest after giving birth

Exclusion Criteria:

* Women who do not want to breastfeed
* Women who have a disability to breastfeed
* Expressing that they cannot continue to work until the end,
* Women who did not participate and did not answer the post-test of the questionnaires.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-26 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Increasing mothers' "breastfeeding self-efficacy scale score" | 12 weeks
  increase in breastfeeding success of lactating puerperant women (After the solution-oriented approach application, the breastfeeding self-efficacy scale The Breastfeeding Self-Efficacy Short Form Scale is a 5-point Likert-Type scale with 1= "I am not sure at all" and 5 = "I am always sure". As Bandura (1998) suggested, all items are positive. The minimum score that can be obtained from the scale is 14, and the maximum is 70.
Increasing "Latch breastfeeding scale score" | 12 weeks
  After the solution-oriented approach application, the latch breastfeeding scale will be evaluated. Each item is evaluated between 0-2 points. The total score that can be taken from the scale is 10. The measurement tool has no cut-off point and the higher the LATCH score, the higher the success of breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: özlem CAGAN, PHD, Principal Investigator — ocagan@ogu.edu.tr
Locations (1):
- Eskisehir Osmnagazi Universty, Eskişehir, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the research results are analyzed and published, access can be made.
Supporting Information: SAP, ICF
Time Frame: 10.08.2023-10.08.2024
Access Criteria: Anyone who works in a similar field, who is interested in this field